CLINICAL TRIAL: NCT05661097
Title: Clinical Study of Hernia Ring Closure Method in Laparoscopic Abdominal Wall Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bo Li (Other)
Responsible Party: Sponsor-Investigator, Bo Li, Chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022006
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Wall Hernia
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Intervention Model Description: random control trail
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Small hernia ring group with continuous suture (Active Comparator): Continuous suture of hernia ring with barbed wire<3cm
  Interventions: Procedure: Suture mode
- Small hernia ring group with discontinuous full-thickness suture (Active Comparator): Intermittent full layer suture to close hernia rings<3cm
  Interventions: Procedure: Suture mode
- Large hernia ring group with continuous suture (Active Comparator): Continuous suture of hernia ring with barbed wire>3cm
  Interventions: Procedure: Suture mode
- Large hernia ring group with discontinuous full-thickness suture (Active Comparator): Intermittent full layer suture to close hernia rings>3cm
  Interventions: Procedure: Suture mode
- Large hernia ring group with continuous suture and discontinuous full-thickness suture (Experimental): Continuous suture with barbed thread and discontinuous full-thickness suture to close hernia rings>3cm
  Interventions: Procedure: Suture mode

INTERVENTIONS:
Procedure: Suture mode — Patients in the small hernia ring group received continuous suture with barbed wire according to simple random method Closure mode, intermittent full layer suture by hernia hook needle.Patients in the large hernia ring group received continuous suture with barbed wire according to simple random method Closure mode, intermittent full layer suture with hernia hook needle, continuous suture with barbed wire+hernia Intermittent full layer crochet suture.

SUMMARY:
By comparing the time of closing the hernia ring, the degree of pain, and the recovery of gastrointestinal tract in different groups Intervening, infection, recurrence and medical cost, to find out whether patients with abdominal wall hernia have different hernias It is the best way to close the hernia ring under laparoscopy and provide evidence based medicine. with In the research process of the research group, a database on abdominal wall hernia will be established for the future Further study of hernia has laid a solid foundation.

ELIGIBILITY:
Inclusion Criteria:

* Conform to the diagnostic criteria of abdominal wall hernia;

  * Patients with general physical condition and can tolerate general anesthesia and laparoscopic surgery; ③ After explaining the situation to the patients and their families, they agreed to join the research group.

Exclusion Criteria:

* The diagnostic criteria of abdominal wall hernia were not met; ② Patients who have serious medical diseases and cannot tolerate laparoscopic surgery; ③ Patients with mental illness; ④ The judgment is affected by incomplete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
recrudescence | 24 months after operation
  Whether abdominal wall hernia recurred within 24 months

SECONDARY OUTCOMES:
Time to close the hernia ring | during operation
  Time to close the hernia ring during operation
Bleeding volume | during operation
  Intraoperative bleeding
Pain level | immediately after the surgery
  Postoperative pain level
Gastrointestinal recovery time | immediately after the surgery
  Postoperative gastrointestinal recovery time
Seroma | immediately after the surgery
  Whether there is seroma after operation
Infected | immediately after the surgery
  Postoperative infection

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfo Mountain Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No